CLINICAL TRIAL: NCT07372833
Title: Natural History Data of International Subjects With an ULTRA-Rare Neuro Developmental Disorder as Part of the ENCORE Expert Clinics, Specifically CAMK2A, CAMK2B, CAMK2D, and CAMK2G.
Brief Title: CAMK2-related Synapthopathies Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Danielle C.M. Veenma, Assistant professor, MD PhD, Erasmus Medical Center
Other Study IDs: MEC-2021-0099
Record Dates: First submitted 2024-11-14; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: CAMK2; Calcium/Calmodulin-dependent Protein Kinase 2
Keywords: CAMK2; Calcium/calmodulin-dependent protein kinase 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biobank for induced pleuripotent stem cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAMK2 mutation: Patients with a mutation in the CAMK2A, CAMK2B, CAMK2D and CAMK2G gene.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without interventions.

SUMMARY:
The key endpoint for this prospective cohort study is:

Mapping of the disease course of all known patients (both children and adults, international) with a CAMK2 mutation, for which ENCORE has founded an expert clinic, and therefore has a substantial and active neuroscientific research arm combined with tertiary academic clinical care delivery for those living in the Netherlands.

Such robust clinical maps can subsequently be used for genotype-phenotype correlations and, identify clinically relevant outcome measures for prognostication, improvement of care delivery & future clinical trials. Additionally, it will most likely generate new research questions for basic scientists who are trying to unravel the specific mechanisms of disease pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a (likely) pathogenic variation in one of the CAMK2 genes
* Consent for anonymous registration in an (inter)national database

Exclusion Criteria:

- Subjects with a Variant of Unknown Significance (VUS); in those cases functional analysis should be performed first.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National and international children and adults with a (likely) pathogenic variation in one of the CAMK2 genes.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2040-01-01 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Age of milestone achievement | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years.
  The TAND (Tuberous Sclerosis Associated Neuropsychiatric Disorders) Checklist collects information on the age at which developmental milestones were achieved, enabling the creation of CAMK2-specific developmental curves.
Presence of seizures | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  Presence of seizures is evaluated through our General questionnaire, which inquires about the presence of comorbidities, and through the online medical interview.
Adaptive Behavior Assessment System 3 (ABAS-3) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The General Adaptive Composite (GAC) score of the ABAS-3 provides an overall estimate of adaptive functioning. Additionally, scores on the different subdomains of the ABAS-3 can be compared with developmental age. The questionnaire consists of 10 subdomains, each with a minimum score of 0 and a maximum score ranging from 66 to 78. Higher scores indicate higher developmental levels.
Social Responsiveness Scale, Second Edition (SRS-2) total score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The SRS-2 measures the severity of social impairment associated with autism spectrum disorder, as individuals with CAMK2-related disorder often exhibit autism spectrum traits. The score from this questionnaire ranges from 0 - 195. For school-aged individuals, scores of 57 and lower are considered to be within normal limits, for pre-school-aged individuals scores of 66 and lower are considered to be within normal limits. Higher scores indicate higher deficiencies in reciprocal social behavior.
Aberrant Behavior Checklist (ABC) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The Aberrant Behavior Checklist measures problem behaviors in individuals with intellectual and developmental disabilities. Scores range from 0 - 174, with higher scores indicating more overall behavioral challenges.

SECONDARY OUTCOMES:
Repetitive Behaviors Questionnaire (RBQ) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The RBQ measures restricted and repetitive behaviors. Scores range from 0 - 76, with higher scores indicating higher frequency of restricted and repetitive behavior.
Child Behavior Checklist (CBCL) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The CBCL measures emotional and behavioral problems. The questionnaire assesses internalizing problems, externalizing problems, and other problems. For children aged 1.5-5 years, scores for internalizing problems range from 0-72, scores for externalizing problems range from 0-48, and scores for other problems range from 0-14. For the 6-18-year-old group, scores for internalizing problems range from 0-64, for externalizing problems from 0-70, and for other problems from 0-72. Higher scores indicate greater problems in these domains.
Children's Behavior Questionnaire (CBQ) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The Children's Behavior Questionnaire (CBQ) measures temperament in early childhood. Subdomains consist of presence of self-injury, severity of self-injury, physical aggression, destruction of property and stereotyped behaviors. Scores range from 0 - 18, with higher scores indicating higher severity of problems.
Mood, Interests and Pleasure Questionnaire Long form (MIPQ-L) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The Mood, Interests and Pleasure Questionnaire monitors emotional well-being and quality of life through subscale scores of mood, interest and pleasure. Scores range from 0-100, with higher scores indicating more positive mood, interest, and pleasure
Short Sensory Profile (SSP) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The Short Sensory Profile questionnaire measures sensory processing patterns. Scores range from 0 - 185, with lower scores indicate more frequent sensory processing difficulties.
Sleep questionnaire for children with neurological andother complex illnesses (SNAKE) score | At baseline and again at the following key developmental ages that have not yet been reached: 3-4 years, 6-7 years, 11-12 years, and 15-17 years. After age 18 years, assessments are repeated every 5 years.
  The SNAKE questionnaire for children with severe psychomotor impairments measures sleep problems in children with severe neurological or psychomotor disabilities. Scores range from 23 - 92, with higher scores indicating more frequent and/or more severe sleep disturbances.
Presence of loss of skills | Assessment with this questionnaire begins at ages 15-17 and is repeated every five years thereafter.
  The LOST-skill questionnaire inquiries about skills in all areas of development and functioning, and stability of body functions, in order to identify patterns of skill loss. Scoring is not used in this questionnaire, as the questionnaire aims to identify patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle CM Veenma, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at the moment